CLINICAL TRIAL: NCT00722150
Title: Artemisinin Resistance in Cambodia II
Acronym: ARC II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Collaborators: World Health Organization (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Mark Fukuda, M.D., LTC, MC, Armed Forces Research Institute of Medical Sciences (AFRIMS)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRAIR 1396; HSRRB number A-14479; WHO RPC252
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Falciparum Malaria
Keywords: Artesunate; Plasmodium Falciparum; Cambodia
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Active Comparator): Oral Artesunate ("standard" dose)
  Interventions: Drug: Artesunate
- Arm 2 (Active Comparator): Oral Artesunate ("ARC1" dose)
  Interventions: Drug: Artesunate
- Arm 3 (Experimental): Oral Artesunate (experimental "high" dose)
  Interventions: Drug: Artesunate

INTERVENTIONS:
Drug: Artesunate — 2 mg/kg/day x 7 days
  Arms: Arm 1
Drug: Artesunate — 4 mg/kg/day x 7 days
  Arms: Arm 2
Drug: Artesunate — 6 mg/kg/day x 7 days
  Arms: Arm 3

SUMMARY:
The purpose of this study is to determine the impact of varying doses of artesunate on treatment outcome and whether higher doses of artesunate can overcome the problem of compromised artemisinin sensitivity in the region.

To determine the safety and tolerability of this previously untested experimental high dose (6 mg/Kg/D X 7 day, total 42 mg/Kg) artesunate monotherapy regimen.

DETAILED DESCRIPTION:
A total of 150 volunteers with acute uncomplicated falciparum malaria will be randomly assigned one of 3 arms to be treated with artesunate monotherapy for 7 days at a ratio of 2:1:2.

Arm 2 serves as a control and will serve as a bridge to the ARC 1 study performed in 2006/2007. Patients in Arm 1 will receive a relatively low "standard" dose, and patients in Arm 2 will receive the intermediate dose of 4 mg/kg that was used in the ARC1 study. Patients in Arm 3 will receive an experimental "high-dose" regimen. Currently available safety data extends to subjects who have received the 28 mg/Kg total dose over 7 days and to another study administering 8 mg/Kg/day for 3 days (total dose 24 mg/Kg). Subjects randomized into this study's 'high-dose' Arm 3 will, therefore, receive a total dose that is higher than has been previously studied in humans.

The study design will be based on the WHO recommendations for the 'Assessment and Monitoring of Antimalarial Drug Efficacy for the Treatment of Uncomplicated Falciparum Malaria' (WHO, 2003).

ELIGIBILITY:
Inclusion Criteria:

1. Acute symptomatic falciparum malaria infection as determined by malaria smear with a parasite density of 1000 to 200,000 asexual parasites/Micro-liter as determined on the thick/thin screening smear with fever (defined as ≥ 37.5ºC), or reported history of fever within the last 48 hours.
2. Age: 18-65 years old
3. All females between the age of 18 and 50 are required to have a negative human chorionic gonadotropin (hCG) pregnancy test (urine). All females of childbearing potential (not surgically sterile, or less than two years menopausal) are required to use an acceptable method of contraception, such as implant, injectable, or oral contraceptive(s), if possible with additional barrier contraception, intrauterine device, sexual abstinence, or vasectomized partner, throughout the study.
4. Written informed consent obtained
5. Willing to stay under close medical supervision for the study duration of 42 days
6. Otherwise healthy Out-patients

Exclusion Criteria:

1. Pregnant women, nursing mothers, or women of childbearing potential who do not use an acceptable method of contraception (as described in Inclusion Criteria, # 3)
2. Mixed malaria infection on admission by malaria smear
3. A previous history of intolerance or hypersensitivity to the study drug artesunate or to drugs with similar chemical structures, such as artemether, artemisinin or dihydroartemisinin
4. History of malaria drug therapy administered in the past 30 days
5. Previous participation in this trial, or participation in any other studies involving investigational or marketed products, concomitantly or within 30 days prior to entry in the study
6. History of significant cardiovascular, liver or renal functional abnormality or any other clinically significant illness, which in the opinion of the investigator would place them at increased risk.
7. Symptoms of severe vomiting (no food or inability to take food during the previous 8 hours).
8. Signs or symptoms of severe malaria (adapted from WHO recommendations (2003): prostration, impaired consciousness, respiratory distress, convulsions, systolic blood pressure < 70 mm Hg, abnormal bleeding, severe anemia with hemoglobin < 8 g/dL or HCT < 24%, hyperparasitemia at > 4% parasitized red blood cells).
9. Unable and/or unlikely to comprehend and/or follow the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Primary clinical outcome is cure (Adequate Clinical and Parasitological Response - ACPR as defined by WHO criteria) on Day 28 and 42 | Day 28 and 42
Safety and tolerability of oral artesunate | Up to 42 days

SECONDARY OUTCOMES:
Secondary outcome measures are time until parasite, fever, and gametocyte clearance (PCT, FCT, and GCT). | Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Delia Bethell, BM BCh, Principal Investigator — Armed Forces Research Institute of Medical Sciences (AFRIMS); Socheat Duong, M.D., Principal Investigator — National Center for Parasitology, Entomology and Malaria Control; Se Youry, M.D., M.P.H.M., Principal Investigator — Armed Forces Research Institute of Medical Sciences (AFRIMS)
Locations (1):
- Tasanh Health Center, Sam Lot District, Battambang, Cambodia

REFERENCES:
- [Derived] Bethell D, Se Y, Lon C, Tyner S, Saunders D, Sriwichai S, Darapiseth S, Teja-Isavadharm P, Khemawoot P, Schaecher K, Ruttvisutinunt W, Lin J, Kuntawungin W, Gosi P, Timmermans A, Smith B, Socheat D, Fukuda MM. Artesunate dose escalation for the treatment of uncomplicated malaria in a region of reported artemisinin resistance: a randomized clinical trial. PLoS One. 2011;6(5):e19283. doi: 10.1371/journal.pone.0019283. Epub 2011 May 13. PMID 21603629
- [Derived] Bethell D, Se Y, Lon C, Socheat D, Saunders D, Teja-Isavadharm P, Khemawoot P, Darapiseth S, Lin J, Sriwichai S, Kuntawungin W, Surasri S, Lee SJ, Sarim S, Tyner S, Smith B, Fukuda MM. Dose-dependent risk of neutropenia after 7-day courses of artesunate monotherapy in Cambodian patients with acute Plasmodium falciparum malaria. Clin Infect Dis. 2010 Dec 15;51(12):e105-14. doi: 10.1086/657402. Epub 2010 Nov 11. PMID 21070142